CLINICAL TRIAL: NCT06843759
Title: Effectiveness of Pilates Exercises Applied to Violinists With Nonspecific Neck Pain : Randomized Controlled Trial
Brief Title: Effectiveness of Pilates Exercises Applied to Violinists With Nonspecific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar21
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Occupational Diseases
Keywords: violinist
MeSH Terms: conditions — Occupational Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mat exercise group (Experimental): mat execises
  Interventions: Other: mat pilates
- reformer exercise group (Experimental): reformer exercises
  Interventions: Other: reformer pilates

INTERVENTIONS:
Other: mat pilates — Neck exercises Trunk stabilization exercises Shoulder exercises Posture exercises
  Arms: mat exercise group
Other: reformer pilates — Foodwork Swan Short Spin Long Stretch Keen Stretch Hug Tree Bridge Pulling Straps Short Box Abdominal Hundred Twist Star
  Arms: reformer exercise group

SUMMARY:
The aim of this study is to examine the effects of different Pilates exercises on violinists experiencing non-specific neck pain

DETAILED DESCRIPTION:
This study is planned as a randomized controlled study. Participants will be divided into two groups, mat pilates and reformer pilates, between the ages of 18-50. Participants will be asked to do the specified exercises for 6 weeks, 2 days a week and 45 minutes each session. Individuals with psychological and physical disabilities to do regular exercise will not be included in the study. The researcher will prepare a personal information form to collect the sociodemographic characteristics of the participants. A visual analog scale will be used to measure pain intensity and recovery process, a neck pain and disability scale to evaluate neck function and disability status, and a neck disability questionnaire to determine the effect of neck pain on daily life activities. These questionnaires will be repeated at the beginning and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-50
* Individuals who play the violin with neck pain
* Having received professional instrument training

Exclusion Criteria

* Using medication
* Having any pathology that prevents exercise
* Having previously undergone upper extremity surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
  Pittsburgh Sleep Quality Index; It evaluates sleep duration, sleep disturbance, sleep efficiency, subjective sleep quality, sleep medication use, daytime dysfunction, and sleep delay and consists of a total of 24 questions. 19 of them are self-report scales and 5 of them consist of questions to be answered by a friend or spouse. There are 7 components with 18 questions scored in the scale, and each component is evaluated between 0 and 3 points. The total score ranges from 0 to 21, and 5 or more is an indicator of "poor sleep quality"
Neck Pain Disability Index Questionnaire | 8 weeks
  The scale includes 10 titles. It includes pain sensitivity, heavy lifting, personal hygiene, reading, sleep, headache, concentration, work, driving, social activities. There are 6 answer options according to the severity of the limitation or pain. Scoring is between 0 and 5. The highest score is 50 and the least is 0. The neck disability level classification according to the total score is as follows 0-4: no restrictions 5-14: mild limitation 15-24: moderate limitation 25-34: severe limitation 34 and up: completely restricted
Bournemouth Neck Pain Survey | 8 weeks
  The survey consists of 7 questions. In addition to questions about pain and disability, it also includes questions about psychosocial issues. Each question is scored between 0 and 10. The highest score is 70, with a higher score indicating a higher level of disability. The content of the survey consists of variables that must be questioned for individuals with neck pain, such as pain severity, the effect of pain on daily life activities and social life, anxiety-depression level, kinesiophobia and coping with pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye Postacı, Study Chair — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steinmetz A, Claus A, Hodges PW, Jull GA. Neck muscle function in violinists/violists with and without neck pain. Clin Rheumatol. 2016 Apr;35(4):1045-51. doi: 10.1007/s10067-015-3000-4. Epub 2015 Jul 15. PMID 26175099
- [Background] Prada V, Mori L, Prato E, Hamedani M, Accogli S, Grandis M, Schenone A. Comparison of Strength and Dexterity in Professional and Student Violinists: Setting Foundations to Guide Rehabilitation. Med Probl Perform Art. 2020 Sep;35(3):130-137. doi: 10.21091/mppa.2020.3021. PMID 32870964
- [Background] Kuo YL, Lee TH, Tsai YJ. Evaluation of a Cervical Stabilization Exercise Program for Pain, Disability, and Physical Impairments in University Violinists with Nonspecific Neck Pain. Int J Environ Res Public Health. 2020 Jul 28;17(15):5430. doi: 10.3390/ijerph17155430. PMID 32731521
- [Background] Chi JY, Halaki M, Ackermann BJ. Ergonomics in violin and piano playing: A systematic review. Appl Ergon. 2020 Oct;88:103143. doi: 10.1016/j.apergo.2020.103143. Epub 2020 May 22. PMID 32678769